CLINICAL TRIAL: NCT05648942
Title: Can Pre-operative Anemia be Timely Identified and Optimized in Patients Awaiting Primary Arthroplasty Surgery? A Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Blood Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200795-01H
Record Dates: First submitted 2022-11-23; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Anemia; Hip Osteoarthritis
MeSH Terms: conditions — Anemia; Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - anemia testing (Experimental): All patients in the experimental group will undergo a point of care test. Patients who meet the higher point-of-care-testing thresholds as possibly having anemia (female: 130g/L; male: 140g/L) will have a formal complete blood count (CBC) test. Formal CBC will not be ordered for all patients in the experimental group to limit the burden on hospital resources. The study co-ordinator will review CBC levels and contact patients to inform them of their results. Patients identified as having anemia in the formal CBC test will be invited to be reviewed in the PBOC.
  Patients in the experimental group who do not meet the threshold for possible anemia on the point-of-care test will continue the current pathway and be reassessed in the preoperative assessment clinic at the time of scheduled surgery. Patients in the experimental group who are determined not to have anemia after formal CBC tests will follow the same pathway.
  Interventions: Diagnostic Test: Anemia testing
- Control (No Intervention): Patients in the control group will not be tested at point of care and will continue on the current pathway and be assessed in the preoperative assessment clinic at the time of scheduled surgery.

INTERVENTIONS:
Diagnostic Test: Anemia testing — Patients will undergo a point of care test to identify possible anemia
  Arms: Experimental - anemia testing

SUMMARY:
Reducing the occurrence of anemia (low circulating hemoglobin levels) post-surgery has been associated with improved outcome, as it reduces complications and allows for faster return to pre-operative function. Post-operative hemoglobin level is dependent upon its pre-operative value (for a given amount of blood loss). About 17% of patients at the Ottawa Hospital (TOH), will be anemic pre-operatively, and if left untreated the patients will have significantly inferior outcomes compared to non-anemic patients. In order to improve outcomes, when a patient is identified as anemic, typically at the pre-operative assessment clinic, he/she is invited to be reviewed and optimized at the Pre-operative Blood Optimization Clinic (PBOC). However, only a quarter of anemic patients are seen in the PBOC due to the lack of time available between anemia identification and surgery and the current resources available. This project will focus on hemoglobin level optimization of pre-operative hip and knee, primary, arthroplasty patients to demonstrate whether early assessment and treatment of pre-operative anemia can be successfully integrated into practice and its impact on post-operative outcomes. Patients will be randomly assigned to either the current standard of care pathway with an anemia test at the pre-operative assessment clinic (2-4 weeks before surgery), at which time they have the option to seek treatment. Patients who are randomly selected to be in the experimental group, will undergo a test to detect anemia at the time they consent for surgery, which is usually 4-6 months prior to surgery. Patients with anemia, will be invited for treatment at the blood optimization clinic at this time. In doing so, this project will test whether timely identification and simple measures is feasible and whether such practice can reduce the overall anemia burden and ultimately improve patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Undergoing primary arthroplasty procedure
* Willing and able to provide informed consent

Exclusion Criteria:

* Patients who are not eligible for assessment and optimization in the preoperative blood optimization clinic. This includes patients with end-stage renal disease (ESRD) or other renal conditions under the care of nephrologists, receiving erythropoietin treatment
* Patients with known hematological malignancy or other hematological conditions which are already on some form of anemia treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Enrollment | Two years
  Number of participants enrolled and willingness of participants to be randomized Comparing the Number of patients screened compared to the number of patients meeting eligibility criteria.
  Tracking crossover between the treatment groups, participant retention, and follow-up rates.
Study Feasibility - Follow-up | Two years
  Rates of participant follow-up
Compliance with treatment in the experimental arm | two years
  Number of participants who complete treatment in the experimental arm
Commencement of treatment by family doctor or self-medication by patients in control arm | two years
  Number of control patients who begin treatment for anemia through family physician or self-medication

SECONDARY OUTCOMES:
Hemoglobin levels | two years
  Hemoglobin levels of both groups at the time of arthroplasty as measured at the pre-operative assessment clinic
Change in hemoglobin | two years
  Change in hemoglobin level in the experimental arm between first formal assessment and pre-operative assessment clinic
Anemia prevelence | two years
  Prevalence of anemia at the time of arthroplasty procedure

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No